CLINICAL TRIAL: NCT05636982
Title: Effectiveness of a Telecare-based Intervention Programme in Supporting the Informal Caregivers of Community-dwelling Older Adults in Reducing Stress Level: Study Protocol for a Pilot Randomized Controlled Trial
Brief Title: A Telecare-based Intervention in Reducing Stress Level of Informal Caregivers of Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Principal investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P0038343
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Telemedicine
Keywords: telecare; older adults; informal caregivers; community

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telecare-based intervention program (Experimental): This group of participants will receive a 3-month telecare-based intervention program which includes three main components: 1) online nurse case management supported by a health-social partnership team, 2) individual-specific video messages covering caregiving skills via WhatsApp, and 3) online information center and discussion forum via a password-protected, newly-developed caregiver website.
  Interventions: Other: Telecare-based intervention program
- Control (No Intervention): The control group will receive conventional community services. The caregiver will attend five educational sessions that covers caregiving skills in the community centers on a fixed schedule.

INTERVENTIONS:
Other: Telecare-based intervention program — A 3-month telecare-based intervention program
  Arms: Telecare-based intervention program

SUMMARY:
The primary caregivers of older adults provide intimate and immediate support when their loved one is in urgent need. Due to the full-time commitment in a caregiving role, the caregiver may not have extra time to join the onsite community services that are available to them in the daytime. With the support of advanced technology, telecare seems to be a convenient and easily accessible channel to provide individualized caregiving advice to the caregivers. This study examines the effectiveness of a telecare-based intervention programme for caregivers.

DETAILED DESCRIPTION:
Objectives: The primary caregivers of older adults provide intimate and immediate support when their loved one is in urgent need. Due to the full-time commitment in a caregiving role, the caregiver may not have extra time to join the onsite community services that are available to them in the daytime. With the support of advanced technology, telecare seems to be a convenient and easily accessible channel to provide individualized caregiving advice to the caregivers. This study examines the effectiveness of a telecare-based intervention programme for caregivers.

Hypothesis to be tested: To test if the research team-developed telecare-based intervention programme is effective in reducing the stress level of caregivers.

Design and subjects: This is a single-blinded, two-armed pilot randomized controlled trial. The subjects are people who are aged 18 or above, provide care to older adults aged ≥ 60 at least 4 hours per week for a minimum of 3 months, are capable to use smartphone to access the Internet, and are without psychiatric illnesses and cognitive impairment.

Interventions: The intervention group receives the telecare intervention programme designed by the research team. The caregivers receive nurse case management supported by a community health-social service team and be able to access a peer-support discussion forum. The control group receives usual community services

Primary outcome measure: Self-reported stress level; secondary outcome measures: self-efficacy, depression level, quality of life, and caregiving burden.

Data analysis: independent t-test or Mann-Whitney U test will be used to determine the group differences in outcomes measurements between pre- and post-intervention. Intention-to-treat will be employed as the primary analysis in this study. Per-protocol (PP) analysis will be adopted as the secondary analysis and performed separately.

Expected outcomes: Caregivers in the intervention group would benefit from the telecare-based programme with reduced stress level, depression level and caregiving burdens and yet enhanced self-efficacy and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* people who are aged ≥18 years old
* understand and communicate in Cantonese
* provide care to the older adults aged ≥60 at least 4 hours per week for a minimum of 3 months
* smartphone user and know how to access the Internet
* commit to attend bi-weekly, 15-30mins online meetings with the program providers over the 3-month period
* willing to receive individual-specific video messages covering caregiving skills via WhatsApp

Exclusion Criteria:

* alcoholic drinkers or psychiatric drug users
* illiterate (inability to write and read)
* having psychiatric problems
* having cognitive impairment as evidenced by scoring 22 or above in Hong Kong version of Montreal Cognitive Assessment
* already participated in other telecare health or social programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Stress level | 3-month
  Stress level will be measured by the 14-item Chinese version of Perceived Stress Scale (PSS). It has been applied extensively to measure the degree of perceived stress for informal caregivers. The total score ranges between 0 (minimum stress perceived) and 56 (maximum stress perceived), with a higher score representing a greater perceived stress level.

SECONDARY OUTCOMES:
Self-efficacy | 3-month
  The General Self-Efficacy Scale (CGSE) will be used to assess the self-perceived ability to cope with stressful life events. The Chinese version of CGSE contains 10 items and is scored on a 4-point Likert scale ranging from 1 (not at all true) to 4 (exactly true). The total score ranges from 10 to 40, with higher scores indicating a greater belief in one's competence to deal with difficulties.
Depression | 3-month
  Depression level will be measured by the Chinese version of The Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a self-reported scale that measures the presence of depressive symptoms. This 4-point scale is a 20-item instrument. The total scores ranged from 0 to 60, with higher scores indicating more depressive symptoms.
Quality of life (general well-being of individual) | 3-month
  The Chinese (HK) version (SF-12v2-HK) of 12-item Short Form Health Survey version 2 will be used to assess the quality of life of the informal caregivers. The questionnaire contains 12 items involving different domains of health concepts, which include physical functioning, role limitation due to emotional problems, role limitation due to physical problems, mental health scale, general health, bodily pain, and social functioning and vitality (energy/fatigue). The scale ranged from 0 to 100, with 50 indicating the standardized norm scale.
Caregiving burden | 3-month
  Caregiving burden will be measured using the Zarit Burden Interview (ZBI). It contains 22 items and is scored on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always). The total score ranges from 0 to 88, with a score of 24 or above may indicate a higher chance of developing depression.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Salvation Army, Kowloon, Hong Kong

REFERENCES:
- [Derived] Wong AKC, Ng NP, Hui VCC, Montayre J. Effect of a telecare-based intervention on stress levels in informal caregivers of older adults: protocol for a randomized controlled trial. Front Psychiatry. 2023 May 25;14:1167479. doi: 10.3389/fpsyt.2023.1167479. eCollection 2023. PMID 37377468